CLINICAL TRIAL: NCT00141505
Title: Placebo-controlled Study on the Pharmacokinetics,Pharmacodynamics, Safety and Tolerability of Concurrent Valproate and Bifeprunox Administration in Subjects With Bipolar I Disorder
Brief Title: PK Effects of Bifeprunox & Valproate in Bipolar I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S154.2.015
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2007-09

CONDITIONS: Bipolar I Disorder
Keywords: drug interaction; pharmacokinetics; valproate; bipolar
MeSH Terms: interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox

SUMMARY:
The study is to evaluate the effect of bifeprunox on the pharmacokinetics of valproate in subjects with Bipolar I Disorder after multiple dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18-65 years old
* meeting DSM-IV criteria for Bipolar I Disorder, either manic or mixed episodes, with or without psychotic features

Exclusion Criteria:

* subjects who are acutely manic, acutely depressed, psychotic or subjects with a current Axis I primary psychiatric diagnosis other than Bipolar I Disorder based on DSM-IV TR criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Atlanta, Georgia, United States